CLINICAL TRIAL: NCT04481165
Title: Subjective Experience of Adolescents Suffering From Anorexia Nervosa With Antidepressants
Brief Title: Experience of Adolescents With Anorexia Nervosa Towards Antidepressants
Acronym: E3A
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200104
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Adolescents Cared for Anorexia Nervosa at Maison de Solenn
Keywords: Anorexia nervosa; Adolescents; Antidepressive agents
MeSH Terms: conditions — Anorexia Nervosa | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adolescents with anorexia nervosa: Adolescents from 12 to 25 year old, cared for anorexia nervosa at the Maison de Solenn (Cochin hospital, Paris, France) et for whom antidepressive agents have been prescribed
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Oral interview and written questions

SUMMARY:
The purpose of this study is to explore the experience of adolescents suffering from anorexia nervosa confronted with the prescription of antidepressants

DETAILED DESCRIPTION:
In our adolescent psychiatric unit, antidepressant's prescription is common during the care pathway for adolescents with anorexia nervosa.

The literature highlights a paradox between scientific data and clinical practice, based on expert consensus. There are a very few qualitative studies in this subject and none of them concern adolescents.

The purpose of this qualitative study is to explore the experience and opinion of adolescents suffering from anorexia nervosa confronted with the prescription of antidepressants

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12 to 25
* Suffering from anorexia nervosa [according to DSM-5 criteria]
* Has been prescribed for a type of SSRIs antidepressant (still ongoing or interrupted at the time of the interview)
* Non-opposition to the study

Exclusion Criteria:

* Atypical eating disorder that do not meet DSM-5 criteria for restrictive anorexia nervosa
* Body Mass Index < 15
* Prescribed for another antidepressant than SSRIs

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescents (between 12 and 25 years) suffer from anorexia nervosa, at the Maison de Solenn, Cochin Hospital, Paris, France
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Qualitative data / Experience of taking anidepressants | At the time of inclusion (Day 0)
  Subjective experience of adolescents with anorexia nervosa about prescription of antidepressants and their effects will be obtained during the grid interview and through their describing to written questions

CONTACTS AND LOCATIONS:
Overall Officials: Maude LUDOT, Psychiatrist, Principal Investigator — APHP, Hôpital Cochin, Maison de Solenn, F-75014 Paris, France; Marie-Rose MORO, PU-PH, Study Chair — APHP, Hôpital Cochin, Maison de Solenn, F-75014 Paris, France; Corinne BLANCHET, PH, Study Director — APHP, Hôpital Cochin, Maison de Solenn, F-75014 Paris, France; Jonathan LACHAL, PHU, Study Director — APHP, Hôpital Cochin, Maison de Solenn, F-75014 Paris, France
Locations (1):
- Maison de Solenn / Cochin Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
* Use of a treatment database, named Actipidos
  * Interview recording on a Dictaphone [kept all over the study in a locked drawer in a medical office at the Maison de Solenn, and then destroyed].
  * Verbatim transcription, on a word-formatted file from a computer in a medical office at the Maison de Solenn; computer secured by a password.
  * Transcripts will be anonymized with an identical number as soon as they are created; no non-anonymized data records will be kept beyond the end of the study.
Supporting Information: Study Protocol, ICF
Time Frame: 6 months after publication
Access Criteria: Interviews will be analysed with a qualitative methodology (Interpretative Phenomenological Analysis)
  - Emergent themes will be presented.

REFERENCES:
- [Background] Leble N, Radon L, Rabot M, Godart N. [Depressive symptoms during anorexia nervosa: State of the art and consequences for an appropriate use of antidepressants]. Encephale. 2017 Feb;43(1):62-68. doi: 10.1016/j.encep.2016.02.017. Epub 2016 Jul 21. French. PMID 27452149
- [Background] Anderson C, Roy T. Patient experiences of taking antidepressants for depression: a secondary qualitative analysis. Res Social Adm Pharm. 2013 Nov-Dec;9(6):884-902. doi: 10.1016/j.sapharm.2012.11.002. Epub 2012 Dec 4. PMID 23219056
- [Background] Ludot-Gregoire M, David V, Carretier E, Lachal J, Moro MR, Blanchet C. Subjective Experience of Antidepressant Prescription Among Adolescents With Anorexia Nervosa. Front Psychiatry. 2022 Apr 4;13:770903. doi: 10.3389/fpsyt.2022.770903. eCollection 2022. PMID 35444576